CLINICAL TRIAL: NCT01890811
Title: Chronic Kidney Disease in Relation to Alterations in Protein and Amino Acid Metabolism and Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-0294
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Failure
Keywords: CKD; Hemodialysis; Protein Digestion; Fat Digestion; Gut Function; Glucose Absorption; Muscle Function
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Boost High Protein (Experimental): Boost high protein with added spirulina
  Interventions: Dietary Supplement: Boost High Protein

INTERVENTIONS:
Dietary Supplement: Boost High Protein — Subjects will receive stable amino acid isotopes IV and will receive Boost High Protein with added isotopes to measure anabolic response to a meal.

SUMMARY:
Weight loss commonly occurs in patients with chronic kidney disease (CKD), negatively influencing their quality of life, treatment response and survival. Loss of muscle protein is generally a central component of weight loss in CKD patients but patients also have reductions in fat mass and bone density, independent of the severity of the disease state. Attempts to reverse weight and muscle loss in CKD and improve nutritional status by nutritional supplementation have been unsuccessful and there are currently no approved therapies.

Purpose of this study is to provide detailed insight in disease related gut function by obtaining information on gut permeability, digestion and absorption of glucose, fat and protein in CKD patients compared to matched healthy controls. Additionally, to examine whether protein and amino acid metabolism is disturbed in CKD patients compared to healthy controls. This will provide required information that will lead to implement new strategies to develop optimal nutritional regimen in order to enhance nutritional status, quality of life and survival in relation to kidney disease.

DETAILED DESCRIPTION:
This study involves one test day of approximately 7-8 hours. On this test day subjects will ingest a sugar drink to assess gut permeability and gut function, and a protein meal to measure digestion/absorption and the anabolic response to food intake. Subjects will also receive a mixture of amino acids that are made a little heavier than normal, called stable isotopes. This stable isotopes is used to investigate protein behavior in the body (protein kinetics). Blood (100-120 ml in total) and urine samples will be collected over 7.5 hours.

ELIGIBILITY:
Inclusion criteria CKD subjects

* Ability to walk, sit down and stand up independently
* Age 55 years or older
* Ability to lie in supine or elevated position for 7 hours
* Diagnosis of kidney disease; undergoing hemodialysis
* Clinically stable condition; no hospitalization 4 weeks preceding first study day
* Willingness and ability to comply with the protocol

Inclusion criteria healthy subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 55 years or older (older control group)
* Ability to lay in supine or elevated position for 7 hours
* No diagnosis of CKD
* Willingness and ability to comply with the protocol

Exclusion Criteria all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (healthy subjects only)
* Established diagnosis of malignancy
* Established diagnosis of Insulin Dependent Diabetes Mellitus
* History of untreated metabolic diseases including hepatic disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Body mass index >40 kg/m2 (healthy subjects only)
* Any other condition that would interfere with the study or safety of the patient (according to the PI or nurse)
* Use of protein or amino acid containing nutritional supplements within 5 days of first study day
* Use of long-term oral corticosteroids or short course of oral corticosteroids within 4 weeks preceding first study day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Net whole-body protein synthesis | 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 min post-meal
  Change in whole-body protein synthesis rate after intake of meal

SECONDARY OUTCOMES:
Citrulline Rate of appearance | Postabsorptive state during 3 hours
  Plasma enrichment of citrulline
Glucose absorption | 7 hours
  Recovery of 3-O-Methyl-D-glucose in the urine.
Gut permeability | 7 hours
  Recovery of rhamnose/lactulose in urine
Skeletal and respiratory muscle strength | 1 day
  Difference in leg strength and fatigue, handgrip strength and fatigue, and inspiratory and expiratory pressure between heart failure patients and healthy controls.
Cognitive function | 1 day
  Outcome of neuro-psychological tests in heart failure patients and healthy controls in relation to the tryptophan metabolism
Fatty acid digestion after feeding | 0,15,30,45,60,75,90,105,120,150,180,210 min post-meal
  Enrichment in palmitic acid and tripalmitin fatty acids in plasma
Protein digestion after feeding | 0,15,30,45,60,75,90,105,120,150,180,210, min post-meal
  Ratio enrichment free phenylalanine vs phenylalanine from protein spirulina
Arginine turnover rate | Postabsorptive state during 3 hours
  Arginine enrichment in plasma
Whole body collagen breakdown rate | Postabsorptive state during 3 hours
  Hydroxyproline enrichment in plasma
Tryptophan turnover rate | Postabsorptive state during 3 hours
  Tryptophan enrichment in plasma
Insulin response to feeding | During 3 hours after feeding
  Acute change from postabsorptive state after intake of meal
Fat-free mass | Postabsorptive state during 15 min
  Characteristics of study subjects
Myofibrillar protein breakdown rate | 0,15,30,45,60,75,90,105,120,150,180,210 min post-meal
  3-Methylhistidine enrichment in plasma
Glycine rate of appearance | Postabsorptive state during 3 hours
  Glycine enrichment in plasma
Taurine turnover rate | Postabsorptive state during 3 hours
  Enrichment of taurine in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University, College Station, Texas, United States